CLINICAL TRIAL: NCT02014415
Title: Alpha-1 Antitrypsin Deficiency Adult Clinical and Genetic Linkage Study
Brief Title: Alpha-1 Antitrypsin Deficiency Adult Liver Study
Status: Active, not recruiting | Type: Observational
Sponsor: St. Louis University (Other)
Collaborators: Alpha-1 Foundation (Other); University of California (Other); Boston University (Other); University College, London (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Jeffrey Teckman M.D., Professor of Pediatrics and Professor of Biochemistry and Molecular Biology, St. Louis University
Other Study IDs: A1F-SLU-7113; Alpha-1 Foundation (Other Grant/Funding Number: A1F-SLU-7113); 22609 (Other: Saint Louis University IRB)
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Alpha-1 Antitrypsin Deficiency
Keywords: Alpha-1; AAT Deficiency; AATD; Liver; Fibrosis; Liver Transplant; Cirrhosis
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples With DNA — Samples of serum, plasma, and blood for genetic testing (Induced Pluripotent Stem Cells (iPS cells), microRNA and DNA) will be collected from subjects at defined time points. In addition, samples of liver tissue will be collected from participants in the Liver Biopsy Group.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Liver Biopsy: Participants will provide liver tissue specimens collected at the time of liver biopsy, to determine the rate of progression of liver injury in adults with Pi-ZZ Alpha-1 Antitrypsin Deficiency.
  Interventions: Procedure: Liver Biopsy (Biopsy Group Only)
- Known Severe Liver Disease: Participants will provide samples of serum, plasma, and DNA at defined time points to determine what genetic and environmental modifiers and biomarkers are associated with severe clinical liver disease, such cirrhosis, portal hypertension and liver failure in adults with Pi-ZZ Alpha-1 Antitrypsin Deficiency.
- Post Liver Transplant: Participants will provide a DNA sample to determine what genetic and environmental modifiers are associated with the need for liver transplantation in adults with Pi-ZZ Alpha-1 Antitrypsin Deficiency.

INTERVENTIONS:
Procedure: Liver Biopsy (Biopsy Group Only) — A percutaneous (needle) liver biopsy will be performed on subjects in the Liver Biopsy Group, in Year 1 and Year 5 of the study.
  Groups: Liver Biopsy

SUMMARY:
The investigators hypothesize that there is liver injury (inflammation, fibrosis, cirrhosis) in adults with Alpha-1 Antitrypsin Deficiency (AATD), which is asymptomatic, under-recognized, and undiagnosed. In addition, the investigators believe that the genetic and environmental factors that play an important role in the development of alpha-1 antitrypsin (AAT) liver disease, can be identified by comparing a cohort database of clinical disease information to linked biospecimen and DNA samples.

DETAILED DESCRIPTION:
Alpha-1 Antitrypsin Deficiency (AATD) is a genetic disorder resulting in a low level of a protein called alpha-1 antitrypsin (AAT). This deficiency can cause life-threatening liver disease and/or lung disease at various ages. Some patients experience life-threatening liver disease in childhood or liver cancer as adults. There is no specific treatment for AAT related liver disease. Some patients develop emphysema as young adults, while some patients remain healthy throughout their lives. Differences in the environment or in other genes may explain such inconsistency in the disease.

The primary objective of this multi-center study is to assess the natural history of individuals with Pi-ZZ AAT deficiency, identify biomarkers for the progression of liver disease and construct a database capable of linking cohort data with repository biospecimens. The secondary objective is to analyze components of the demographic, social, and family history associated with more severe liver disease.

This study will examine the natural history of liver disease by recording participant's family history, medical history, current health, laboratory test results, and medical treatment(s). Participants may complete brief research questionnaires about their physical and mental health, diet, alcohol intake, and smoke, environmental and occupational (work) exposures.

At least 120 Pi-ZZ AAT deficient adults with no previous history of liver disease, moderate-severe liver disease, or post liver transplant, will be enrolled at one of three sites. Eligible subjects will participate in one of the following study arms:

1. Liver Biopsy
2. Known Severe Liver Disease - subjects not meeting Biopsy Group eligibility due to the presence of advanced liver disease
3. Post Liver Transplant - subjects who have previously undergone a liver transplant

At the time of enrollment, each participant will be assigned a unique study identification (ID) number. All participant information recorded and samples collected for the study will be saved by this unique number. All blood, tissue and genetic samples collected will be sent to a secured repository for future retrieval and study. The process of coding data and samples lessens the chances of a breach in confidentiality.

The length of study participation, tests and activities performed specifically for research will be determined by the enrollment group. Subjects in the Biopsy and Known Severe Liver Disease groups participate in the study for 5 years (enrollment and four annual follow-up visits). Both groups undergo a physical exam, diagnostic abdominal ultrasound, pulmonary function testing and the collection of serum, plasma and blood for routine laboratory and genetic testing (Induced Pluripotent Stem Cells (iPS cells), microRNA and DNA). However, only the Biopsy Group participants undergo a liver biopsy and FibroScan at enrollment, and again in Year 5. The liver tissue samples will help the researchers learn what causes liver disease in some patients and how the liver disease progresses.

Subjects in the Post Liver Transplant group have a single study visit to record their history, complete questionnaires and perform pulmonary function testing. In addition, whole blood for DNA analysis will be collected from these participants.

Based on their study arm assignment, participants will receive copies of their diagnostic abdominal ultrasound, pulmonary function test, routine laboratory test and liver biopsy pathology results, to share with their primary care physician.

Upon completion of the 5-year study, two cross-sectional visits were added to the Biopsy Group and Known Severe Liver Disease Group. The cross-sectional visit will be completed by phone and review of medical records.

ELIGIBILITY:
Liver Biopsy Group:

Inclusion Criteria

* Adults (≥ 18 years of age), with Alpha-1 Antitrypsin Deficiency
* Documented evidence Pi-ZZ phenotype or genotype
* Both genders, all races and ethnic groups
* Willingness to be followed for up to 5 years

Exclusion Criteria:

* Evidence of advanced liver disease defined by Child-Pugh Class B or C (score ≥ 7)
* Known advanced lung disease defined as forced expiratory volume at one second (FEV1) < 40 % of Predicted
* History of Organ Transplantation
* Known congenital or metabolic liver disease (e.g.: Wilson's, glycogen storage, cystic fibrosis)or iron overload as evidenced by ≥ Grade 3 iron staining on a previous liver biopsy
* Evidence of chronic hepatitis B (marked by the presence of HBsAg in serum) or Hepatitis C (marked by the presence of anti-hepatitis C virus (HCV) or HCV RNA in serum)
* Vascular disorders of the liver (e.g.: cardiac sclerosis, acute or chronic Budd-Chiari, hepatoportal sclerosis, peliosis)
* Known HIV positivity
* Diagnosis of malignancy within the last 5 years
* Active substance abuse, that in the opinion of the study investigator, would interfere with adherence to study requirements
* Concomitant severe underlying systemic illness or medical condition which in the opinion of the investigator, would make the patient unsuitable for the study or would interfere with completion of follow-up
* Inability to comply with the longitudinal follow-up as outlined in the protocol
* Failure of the participant to sign informed consent or Health Insurance Portability and Accountability Act (HIPAA) documents

Known Severe Liver Disease Group:

Inclusion Criteria

* Adults (≥ 18 years of age), with alpha-1-antitrypsin deficiency
* Documented evidence PI-ZZ phenotype or genotype
* Documented evidence of portal hypertension or evidence of advanced liver disease defined by Child-Pugh Class B or C (score ≥ 7), or previous liver biopsy with an Ishak Fibrosis Score ≥ 4
* Both genders, all races and ethnic groups
* Willingness to be followed for up to 5 years

Exclusion Criteria

* History of Organ Transplantation
* Known congenital or metabolic liver disease (e.g.: Wilson's, glycogen storage, cystic fibrosis) and iron overload as evidenced by ≥ Grade 3 iron staining on a previous liver biopsy
* Evidence of chronic hepatitis B (marked by the presence of HBsAg in serum) or Hepatitis C (marked by the presence of anti-HCV or HCV RNA in serum)
* Vascular disorders of the liver (e.g.: cardiac sclerosis, acute or chronic Budd-Chiari, hepatoportal sclerosis, peliosis)
* Known HIV positivity
* Diagnosis of malignancy within the last 5 years which in the opinion of the investigator, would make the patient's follow-up problematic or the results uninterpretable.
* Active substance abuse, that in the opinion of the study investigator, would interfere with adherence to study requirements
* Concomitant severe underlying systemic illness or medical condition which in the opinion of the investigator, would make the patient unsuitable for the study or would interfere with completion of follow-up
* Inability to comply with the longitudinal follow-up as outlined in the protocol
* Failure of the participant to sign informed consent or HIPAA documents.

Post Liver Transplant Group

Inclusion Criteria

* Adults (≥ 18 years of age), with alpha-1-antitrypsin deficiency
* Pre-transplant documented evidence of PI-ZZ phenotype or genotype
* Documented evidence of liver transplantation
* Both genders, all races and ethnic groups

Exclusion Criteria

* Active substance abuse, that in the opinion of the study investigator, would interfere with adherence to study requirements
* Concomitant severe underlying systemic illness or medical condition which in the opinion of the investigator, would make the patient unsuitable for the study or would interfere with completion of study requirements
* Failure of the participant to sign informed consent or HIPAA documents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pi-ZZ AAT deficient adults with either no previous history of liver disease, moderate-severe liver disease or post liver transplant. Biologic family members who are also Pi-ZZ and ≥ 18 years of age, will be offered enrollment into the study. The purpose of including family members is to determine if the natural history of the liver disease is consistent in a given family.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-12; Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The risk and rate of histologic liver injury progression, as measured by liver biopsy, over a 5-year period. | Liver biopsy performed in Year 1 and Year 5

SECONDARY OUTCOMES:
Calculated Model for End-stage Liver Disease score (MELD) | Calculated at baseline and annually through year 5
Liver synthetic dysfunction defined by international normalized ratio (INR) > 1.3 or serum albumin < 3.2 gm/dL | Measured at baseline and annually through year 5
Presence of ascites (or treatment for ascites) | Assessed at baseline and annually through year 5
Development of complications of portal hypertension (e.g., variceal hemorrhage) | Assessed at baseline and annually through year 5
Jaundice (total serum bilirubin >2.0 mg/dl) | Measured at baseline and annually through year 5
Liver transplantation | Assessed annually through year 5
Listing for liver transplantation | Assessed at baseline and annually through year 5
Health related quality of life | Measured at baseline and annually through year 5
FEV1 % of Predicted | Collected at baseline and annually through year 5
Death | Collected annually through year 5

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Teckman, MD, Study Chair — St. Louis University; Andrew A Wilson, MD, Study Director — Alpha-1 Foundation; David A. Brenner, MD, Principal Investigator — The University of California, San Diego; Andrew A Wilson, MD, Principal Investigator — Boston University
Locations (3):
- United States (3):
  - University of California, San Diego, California
  - Boston University School of Medicine, Boston, Massachusetts
  - Saint Louis University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Based on study group assignment, participants will be given a copy of their test results as follows:
  Liver Biopsy Group- liver biopsy pathology, diagnostic abdominal ultrasound, pulmonary function testing, and routine clinical laboratory testing.
  Known Severe Liver Disease Group- diagnostic abdominal ultrasound, pulmonary function testing, and routine clinical laboratory testing.
  Post Liver Transplant Group- pulmonary function testing.